CLINICAL TRIAL: NCT03253211
Title: Disseminating NIH Evidence Based Sickle Cell Recommendations in North Carolina
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: PRO00076048
Record Dates: First submitted 2017-08-02; First posted 2017-08-17 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Sickle Cell Disease
Keywords: Co-management model of care; Primary Care; Specialty Care; Decision support tools; Emergency Department Clinicians; Co-management
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- State: North Carolina
- SCD Patients
- Providers: Primary care and emergency department clinicians
- Year: Baseline, year 2, year 3

SUMMARY:
This project will improve the efficiency and quality of healthcare for persons with sickle cell disease, an under-served and at risk population by implementing a co-management model of care. Many patients with sickle cell disease (SCD) receive care primarily from specialty physicians and emergency departments (ED), thus resulting in a lack of primary care and a high number of ED visits and hospitalizations. The goal is to improve PCP and SCD specialist co-management. The overall purpose of this dissemination project is to evaluate utilization data, as well as patient and provider reported outcomes associated with the dissemination of a toolbox of decision support tools to PCP's and ED providers across NC and SC.

DETAILED DESCRIPTION:
The investigators will achieve the goals stated above through three aims.

1. Examine the effects of decision support tools on study outcomes during the 12 months prior to project start and across the 3.5 years of the project in NC and SC. The investigators will also determine which patient and practice level characteristics predict study outcomes.
2. Evaluate individual provider-reported awareness, use and preference of health maintenance tables and algorithms amongst PCPs and ED providers in NC and SC at project start and yearly across the project. Additionally, the investigators will explore patient reported awareness of and satisfaction with co-management model of care in NC and SC.
3. The investigators will conduct an exploratory cost analysis of the dissemination and implementation of the SCD co-management model and its effect on healthcare resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* patient with diagnosis of sickle cell disease, emergency department clinician, or primary care clinician in the state of NC or part of SC

Exclusion Criteria:

* Non-English speaking, non-resident of NC or SC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of sickle cell disease (not trait) are eligible for inclusion. Additionally, we will survey primary care and emergency department clinicians. Patients must be from North Carolina or Georgetown, SC. Clinicians must practice in NC or SC.
Sampling Method: Non-Probability Sample
Enrollment: 4392 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
HU refills | 12 months
  number of hydroxyurea prescription refills per patient
Co-management visits | 12 months
  number of co-management visits per patient

SECONDARY OUTCOMES:
ED visits | 12 months
  number of visits to the emergency department per patient
In-patient hospitalizations | 12 months
  number of in-patient hospitalizations per patient
Re-admission to hospital within 30 days | 12 months
  number of re-admissions per patient over the course of one year
Primary care visits | 12 months
  number of visits to primary care provider per patient
Specialty visits | 12 months
  number of specialty care visits per patient
Transcranial doppler screening | 12 months
  number of transcranial doppler screenings per patient
Opioid prescription fills | 12 months
  number of opioid prescription fill days per patient

CONTACTS AND LOCATIONS:
Overall Officials: Paula Tanabe, PhD, Principal Investigator — Duke University
Locations (1):
- Community Care of North Carolina, Raleigh, North Carolina, United States